CLINICAL TRIAL: NCT00398463
Title: Tailoring Treatment With Tirofiban in Patients Showing Resistance to Aspirin and/or Resistance to Clopidogrel
Brief Title: Study of Tirofiban Administration in Patients With Aspirin and or Clopidogrel Resistance
Acronym: 3T/2R
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Marco Valgimigli, Azienda Ospedaliera Universitaria di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TCA-01-III
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2008-06

CONDITIONS: Angioplasty, Transluminal, Percutaneous Coronary
Keywords: tirofiban; aspirin resistance; clopidogrel resistance
MeSH Terms: interventions — Tirofiban

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Aspirin, clopidogrel, Unfractioned heparin or bivalirudin plus tirofiban infusion given at high bolus dose
  Interventions: Drug: Tirofiban
- 2 (Placebo Comparator): Aspirin, clopidogrel, Unfractioned heparin or bivalirudin plus placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirofiban — Tirofiban infusion given as high bolus dose plus standard 14-24 hour infusion
  Other Names: Glycoprotein IIb/IIIa inhibitor
  Arms: 1
Drug: Placebo — Saline infusion will be administered for 14-24 hours
  Other Names: Glycoprotein IIb/IIIa inhibitor
  Arms: 2

SUMMARY:
This study will evaluate whether adding tirofiban, administered at high bolus dose on top of aspirin and clopidogrel will lead to a lower rate of periprocedural myocardial infarction after percutaneous coronary intervention in elective patients presenting with aspirin and/or clopidogrel resistance.

DETAILED DESCRIPTION:
This study will investigate the effect of treatment with a high bolus dosage of Tirofiban (in addition to Aspirin, Heparin and 300mg or 600mg clopidogrel) on the rate of periprocedural myocardial infarction compared to Aspirin, Heparin (or bivalirudin) and 300mg or 600mg clopidogrel alone in patients resistant to aspirin and/or to clopidogrel.

This is a randomized, double blind, placebo controlled (with bailout tirofiban as rescue) multicenter study. Enrollment will last between 12 and 36 months depending on the final number of participating centres. The minimum follow-up will be 30 days after the index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. All Patients older than 18 years scheduled for coronary angiography and/or PCI will be enrolled. [Patients should be CK-MB negative (to avoid CK washout with revascularization) and also cTnI/T negative whereas other high-risk features will not lead to patient exclusion.
2. All consecutive patients with stable or unstable troponin and CK-MB negative coronary artery disease showing aspirin and or clopidogrel resistance (ACR) will be enrolled. These include:

   * Patients with clinical indication to undergo angiography for possible revascularisation.
   * Patients with ACR in whom catheter-based coronary intervention is planned based on previous angiogram.

Exclusion Criteria:

1. Patients who can not give informed consent or have a life expectancy of < 1 year
2. Evolving or Ongoing myocardial infarction (MI) (Persistence of or developing Q wave or ST segment elevation at ECG with or without typical chest pain or typical rapid rise and fall CK-MB or new LBBB) or patients in whom the treating physician intends to use a Gp IIB/IIIa inhibitors.
3. Administration of any GP IIb/IIIa receptor antagonist, anticoagulation, or lytic therapy in the previous 30 days
4. Serum creatinine more than 2.5 mg/dl (221 micromol/L)
5. Ongoing bleeding or bleeding diathesis or contraindication for anticoagulation or increase bleeding risk or history of bleeding in the last 1 year
6. Previous stroke or TIA or any intracranial pathology in the last six months
7. Major surgery or trauma within the previous six weeks
8. Platelet count < 100.000 per cubic mm or HCT ,33% or Hb < 11 gm/dL
9. Subjects who received low-molecular-weight heparin within the 24 hours prior to randomization
10. Subjects with an allergy or intolerance to aspirin, heparin, clopidogrel, or tirofiban
11. Patients with severe hypertension (SBP > 180 mm Hg or DBP > 110 mm Hg) or in cardiogenic shock (SBP 80 mm Hg or below for > 30 minutes) or requiring IABP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2006-05; Primary Completion 2008-07 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Troponin I or T elevation ratio at least three times the upper limit of normal. | 48 hours

SECONDARY OUTCOMES:
The incidence of myocardial infarction defined as elevation of CK-MB >1, ≥3 or ≥5 times the ULN in one or more blood sample(s). | 30 days
Elevation of troponin levels above upper limit of normal in ratios different from the primary endpoint | within 30 days
Bleeding rates | 30 days
Stent thrombosis | with the first year of follow-up
The rate of major adverse cardiovascular events | at 30 days and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marco Valgimigli, MD, PhD, Principal Investigator — Università degli Studi di Ferrara
Locations (1):
- Cattedra di Cardiologia, Azienda Ospedaliera Universitaria di Ferrara, Ferrara, Fe, Italy

REFERENCES:
- [Background] Chen WH, Lee PY, Ng W, Tse HF, Lau CP. Aspirin resistance is associated with a high incidence of myonecrosis after non-urgent percutaneous coronary intervention despite clopidogrel pretreatment. J Am Coll Cardiol. 2004 Mar 17;43(6):1122-6. doi: 10.1016/j.jacc.2003.12.034. PMID 15028378
- [Background] Valgimigli M, Percoco G, Barbieri D, Ferrari F, Guardigli G, Parrinello G, Soukhomovskaia O, Ferrari R. The additive value of tirofiban administered with the high-dose bolus in the prevention of ischemic complications during high-risk coronary angioplasty: the ADVANCE Trial. J Am Coll Cardiol. 2004 Jul 7;44(1):14-9. doi: 10.1016/j.jacc.2004.03.042. PMID 15234398
- [Derived] Valgimigli M, Campo G, de Cesare N, Meliga E, Vranckx P, Furgieri A, Angiolillo DJ, Sabate M, Hamon M, Repetto A, Colangelo S, Brugaletta S, Parrinello G, Percoco G, Ferrari R; Tailoring Treatment With Tirofiban in Patients Showing Resistance to Aspirin and/or Resistance to Clopidogrel (3T/2R) Investigators. Intensifying platelet inhibition with tirofiban in poor responders to aspirin, clopidogrel, or both agents undergoing elective coronary intervention: results from the double-blind, prospective, randomized Tailoring Treatment with Tirofiban in Patients Showing Resistance to Aspirin and/or Resistance to Clopidogrel study. Circulation. 2009 Jun 30;119(25):3215-22. doi: 10.1161/CIRCULATIONAHA.108.833236. Epub 2009 Jun 15. PMID 19528337